CLINICAL TRIAL: NCT05971836
Title: The Molecular Basis of Inherited Reproductive Disorders
Status: Recruiting | Type: Observational
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 2020P000762
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hypogonadotropic Hypogonadism; Reproductive Disorder; Kallmann Syndrome; Delayed Puberty
Keywords: Hypogonadotropic hypogonadism; Reproductive disorders; Kallmann syndrome; Kisspeptin; Delayed Puberty
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome; Puberty, Delayed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with Reproductive Disorders: Individuals with reproductive disorders and their affected and unaffected family members

SUMMARY:
The goal of this study is to learn more about the genes that control puberty and reproduction in humans.

DETAILED DESCRIPTION:
All study subjects will undergo the same activities. Subjects will provide up to five tubes of blood for genetic analysis, complete a smell test, and answer questions about their health and family history.

ELIGIBILITY:
Participants must belong to one of the following categories:

* Failure to go through a normal, age-appropriate, spontaneous puberty and low sex steroid levels in the setting of low/normal gonadotropins or,
* Abnormally early development of puberty or,
* Normal puberty with subsequent development of low gonadotropin levels or,
* Evidence of a reproductive disorder with high gonadotropin levels or,
* Pre-pubertal individuals with features suggestive of hypogonadotropic hypogonadism or,
* Affected and unaffected family members of individuals that fit criteria above

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with reproductive disorders and their affected and unaffected family members
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Genetic variation | Day 1
  Identification of one or more genetic variations related to reproductive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No